CLINICAL TRIAL: NCT02372994
Title: My Team of Care (MyTOC) Trial: a Pilot Randomized Controlled Trial of an Online Communication Tool (Loop) for Collaborative Care in Complex Patients
Brief Title: My Team of Care: a Pilot Randomized Controlled Trial of an Online Communication Tool for Collaborative Care
Acronym: Loop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 410001734
Record Dates: First submitted 2015-01-26; First posted 2015-02-26 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Neoplasms; Communication
Keywords: chronic disease; continuity of patient care; patient engagement; cost effectiveness analysis; user-centred design; Interdisciplinary Health Team; Medical Informatics; Patient-centred care
MeSH Terms: conditions — Neoplasms; Communication; Chronic Disease; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): The randomization is at the level of attending healthcare professional who identifies patients for recruitment. For each participant in the intervention arm, a secure space (called a Patient Loop) is created in the online clinical communication system. A Patient Loop can be accessed by the patient, their caregiver, and the healthcare providers who have permission to do so through an algorithm of invitation, authentication and careful partitioning. In each Patient Loop, team members can post messages that can be read and responded to by the entire team. Each Patient Loop consists of a patient, their caregiver and at least two healthcare professionals.
  Interventions: Other: Loop
- Control Group (No Intervention): Participants receive usual care.

INTERVENTIONS:
Other: Loop — Loop is a secure online communication system centered on the patient that assembles the patient's actual healthcare team for ongoing collaborative care. The patient and caregiver are integral members of the team. Loop is cross-organizational, cross-setting and interprofessional. It is for ongoing, interactive, contextual, team-based communication. Loop is explicitly for asynchronous communication, not instant messaging. The stream of messages is stored and can be sorted for ease of viewing. The tool was developed with user-centred design and requires no prior training.
  Other Names: Online Clinical Collaboration System; My Team of Care (MyTOC)
  Arms: Intervention Group

SUMMARY:
This project will pilot and test a new online communication tool, Loop, developed within a research framework with participatory and user-centred design. This pilot trial focuses on advanced cancer as an example of complex care. Cancer care involves many healthcare providers, spanning hospital to home. There is no organized way for them to communicate. Loop is a practical tool for ongoing collaboration in the patient's actual team of care that engages patients. The study will answer the questions: does Loop improve communication efficiency, engage patients and family physicians, and show early benefits in quality and health care costs?

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Stage IV cancer, or Patients with stage III cancer and poor prognosis as determined by a physician (>3 months but <2 years)
2. Eastern Cooperative Oncology Group (ECOG) performance status score ≤2
3. Each patient must have at least two healthcare providers, including an attending oncologist or palliative care physician
4. Patient and, if applicable, family caregiver must be ≥18 years of age
5. Literacy and language capacity and competency to provide informed consent
6. Patient or caregiver must have access to a computer and the internet

Exclusion Criteria:

1. Patients without the capacity to participate in use of the online tool, and do not have a caregiver who can engage in use of the tool on their behalf
2. Participants without the capacity to participate in evaluation of outcome measures, including, but not limited to, online and paper-based multiple-choice questions, checklists, and visual analogue scales, and do not have a family caregiver who can complete outcome measures
3. A potential candidate for or currently receiving hormone therapy for breast or prostate cancer
4. Patients with a prognosis of <3 months as determined by attending physician
5. Patients with impaired mental status as previously assessed by a physician or judged by research staff using the Bedside Confusion Scale
6. It has been determined that the patient is participating in another study precluding them from taking part in this study, as determined by an agreed-upon algorithm, tracked and managed by study coordinators

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Trial feasibility measured with number of patients recruited for study who have consented and participate for the duration of the study. | 1 year

SECONDARY OUTCOMES:
Trial feasibility measured with number of healthcare providers recruited for study who have consented and participate for the duration of the study. | 1 year
Trial feasibility measured with number of family caregivers recruited for study who have consented and participate for the duration of the study. | 1 year
Palliative Care Outcomes Scale | 3 months
  A 12 item questionnaire measuring patient-reported quality of care
Picker Ambulatory Cancer Care Survey Continuity and Coordination subscale | 3 months
  An 8 item questionnaire measuring patient-perceived continuity and coordination of care
Ambulatory and Home Care Record | 3 months
  Measure of ambulatory, home-based and acute care health services utilization, and associated public and private costs
Edmonton Symptom Assessment Scale | 3 months
  A 10 item questionnaire measuring symptom intensity
Eastern Cooperative Oncology Group score | 3 months
  A measure of performance status
The proportion of eligible participants who are invited to participate | 1 year
The proportion of invited participants who consent to participate | 1 year
The mean duration of participation of all study participants | 1 year
Instrument completion rate for the Palliative Care Outcomes Scale | 1 year
Item response rate for the Palliative Care Outcomes Scale | 1 year
Instrument completion rate for the Picker Ambulatory Cancer Care Survey Continuity and Coordination subscale | 1 year
Item response rate for the Picker Ambulatory Cancer Care Survey Continuity and Coordination subscale | 1 year
Instrument completion rate for the Ambulatory and Home Care Record | 1 year
Item response rate for the Ambulatory and Home Care Record | 1 year
Instrument completion rate for the Edmonton Symptom Assessment Scale | 1 year
Item response rate for the Edmonton Symptom Assessment Scale | 1 year
Number of family physicians who participate per study group | 1 year

OTHER OUTCOMES:
Number of posts per participant on the Loop system | 3 months
Number of times a patient logs into the Loop system | 3 months
Number of times a caregiver logs into the Loop system | 3 months
Number of times a healthcare provider logs into the Loop system | At end of study participation
  Healthcare providers will be enrolled in the study for between 3 months and 1 year
Time interval between a message posting by a patient/caregiver and a response by a healthcare provider on the Loop system | 3 months
Number of occurrences of user-reported errors | 3 months
Proportion of functions being used on the Loop system | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Amna Husain, MD MPH, Principal Investigator — Temmy Latner Center for Palliative Care, Mount Sinai Hospital
Locations (2):
- Canada (2):
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Voruganti T, Grunfeld E, Jamieson T, Kurahashi AM, Lokuge B, Krzyzanowska MK, Mamdani M, Moineddin R, Husain A. My Team of Care Study: A Pilot Randomized Controlled Trial of a Web-Based Communication Tool for Collaborative Care in Patients With Advanced Cancer. J Med Internet Res. 2017 Jul 18;19(7):e219. doi: 10.2196/jmir.7421. PMID 28720558